CLINICAL TRIAL: NCT02695667
Title: Quantitative Genioglossal Muscle Strength in Obstructive Sleep Apnea (OSAS) Defined in the Clinical Spectrum of Subjects With Snoring Disturbance, Oral Appliance Therapy Responsive, and CPAP Responsive.
Brief Title: Quantitative Genioglossal Muscle Strength in Obstructive Sleep Apnea (OSAS)
Acronym: EatonOSAS
Status: Terminated | Type: Observational
Why Stopped: This was inadvertently entered in the system and is not a clinical trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 15-120
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSAS subjects: CPAP Referral OSAS
- Risk-Free subjects: paired normal control subjects

SUMMARY:
Quantitative Genioglossal muscle strength in Obstructive Sleep Apnea (OSAS) defined in the clinical spectrum of subjects with Snoring Disturbance, Oral Appliance Therapy Responsive, and CPAP Responsive

DETAILED DESCRIPTION:
To describe by statistical analysis the normal distribution domain of genioglossus muscle strength in each of the four clinical stages of Sleep Apnea; and, by regression analysis, to explore the possibility of an inverse relationship between decreasing genioglossus strength and progression of the clinical stages of OSAS.

1.3. To test the hypothesis that a "subpopulation of subject" exists within the clinical spectrum of OSAS, in whom decreasing strength of the genioglossus muscle may represent a common element in spite of differing possible pathophysiologic pathways leading to Obstructive Sleep Apnea in man. 1.4. The major hypothesis of this proposal is thus that "Genioglossal Strength is inversely correlated with Obstructive Sleep Apnea Pathology."

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years inclusive BMI 18-25 Non-smoking history and no current use for a minimum of 6 months No smokeless tobacco products (including e-cigarettes) for a minimum of 6 months No sleep snoring reported by subject and by bedroom "companion" Self-described as active/athletic (i.e. regular hikes, walks, jogging, running, active Sports, such as volleyball, soccer, etc.) Self-described as healthy, with no known disease or recent illness Self-completed Epworth Sleepiness Scale of <6 (Johns, MW, A new method for Measuring daytime sleepiness: the Epworth Sleepiness Scale; SLEEP 14:450-5, 1991). Physical Examination Mallampati Score of Class 1 (Nuckton, TJ, et al: Physical

Examination: Mallampati Score as an Independent Predictor of OSAS; SLEEP 29:

903-908, 2006).

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This initial pilot investigation will screen up to 70 individuals to obtain the necessary enrollment of 22 subjects per group from Stage Three: CPAP Referral OSAS; and paired normal control subjects
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Genioglossal Strength | single clinic visit
  quantitative measurement of tongue strength

CONTACTS AND LOCATIONS:
Overall Officials: Philip Eaton, MD, Principal Investigator — University of New Mexico
Locations (1):
- Clinical Translational Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No